CLINICAL TRIAL: NCT04077060
Title: First Trimester Risk Assessment Based on Ultrasound and Cell-free DNA vs Combined Screening: Women's Experience
Brief Title: First Trimester Risk Assessment Based on Ultrasound and Cell-free DNA vs Combined Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 209/19
Record Dates: First submitted 2019-08-26; First posted 2019-09-04 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Aneuploidy
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPT (Experimental): Women randomized in the intervention group will be offered cfDNA screening, along with an early detailed anatomy scan, including nuchal measurement, at 11-13 weeks of gestation. cfDNA analysis will include a simultaneous microarray-based assay of non-polymorphic (chromosomes 13, 18, 21, X and Y) and polymorphic loci to estimate chromosome proportion and fetal fraction. NIPT will be performed at the time of randomization or after if gestational age at randomization < 9 6/7 weeks of gestation.
  Interventions: Diagnostic Test: NIPT
- Combined screening (Other): Control group includes the standard of care. In our department, first-trimester risk assessment is performed routinely at 11-13 weeks of gestation by FTCS as per standard of care. FTCS includes crown-rump length, NT measurements, and a detailed ultrasound examination based on ISUOG guidelines. All operators who perform this examination are certified by the UK Fetal Medicine Foundation (FMF). A specific risk for aneuploidy is not calculated if NT measurement is >3.5 mm or if fetal anomaly is identified. These cases are deemed to be at a very high risk for chromosomal abnormalities and are offered invasive testing.
  Interventions: Diagnostic Test: combined screening

INTERVENTIONS:
Diagnostic Test: NIPT — Women randomized in the intervention group will be offered cfDNA screening, along with an early detailed anatomy scan, including nuchal measurement, at 11-13 weeks of gestation. cfDNA analysis will include a simultaneous microarray-based assay of non-polymorphic (chromosomes 13, 18, 21, X and Y) and polymorphic loci to estimate chromosome proportion and fetal fraction. NIPT will be performed at the time of randomization or after if gestational age at randomization < 9 6/7 weeks of gestation.
  Women in both groups will be given oral counseling by obstetricians and will be counseled about test procedures, reporting time, test sensitivity and specificity, and the necessity to confirm abnormal screening results with invasive testing.
  Arms: NIPT
Diagnostic Test: combined screening — Control group includes the standard of care. In our department, first-trimester risk assessment is performed routinely at 11-13 weeks of gestation by FTCS as per standard of care. FTCS includes crown-rump length, NT measurements, and a detailed ultrasound examination based on ISUOG guidelines. All operators who perform this examination are certified by the UK Fetal Medicine Foundation (FMF). A specific risk for aneuploidy is not calculated if NT measurement is >3.5 mm or if fetal anomaly is identified. These cases are deemed to be at a very high risk for chromosomal abnormalities and are offered invasive testing.
  Arms: Combined screening

SUMMARY:
There is an ongoing debate regarding how cell-free DNA (cfDNA) screening can best be incorporated into current prenatal screening algorithms for chromosomal abnormalities.

Test performance of cfDNA has been shown to be better that first-trimester combined screening (FTCS). However, the cost of the cfDNA testing is considered too high to adopt as first line screening. Moreover, FTCS includes a detailed ultrasound examination of the fetus with nuchal translucency (NT) measurement that allows for early detection of fetal abnormalities.

An approach in which every woman are offered an early anatomy scan along with cfDNA may also be a reasonable option. Recently a randomized controlled trial, including 1,518 women with singleton pregnancy undergoing first-trimester screening, compared the screening performance of FTCS with an approach that uses the combination of a detailed ultrasound examination and cfDNA analysis. The trial showed that first-trimester risk assessment for trisomy 21 that includes a detailed ultrasound examination along cfDNA was associated with a significant reduction in the false-positive rate compared with FTCS. This approach obviates the need for maternal serum free beta-human chorionic gonadotropin and pregnancy-associated plasma protein-A in screening for fetal aneuploidy.

Despite robust evidence on the very high detection rate of cfDNA in detecting trisomy 21, literature is lacking on data regarding women's experience and emotional well-being and satisfaction after test-results of women offered cfDNA compared to those offered FTCS.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton gestations
* ≤12 6/7 weeks of gestation
* Normal ultrasound examination at the time of randomization
* >18 <45 years
* Crown-rump length (CRL) <84 mm at the time of randomization

Exclusion Criteria:

* Multiple gestations, including vanishing twins
* >12 6/7 weeks of gestation
* Ectopic pregnancy
* Abnormal ultrasound examination at the time of first prenatal visit
* Women who are unconscious, severly ill, mentally handicapped, or under the age of 18 years.
* Women who have already planned for invasive prenatal testing, e.g. for a history of prior child or pregnancy with chromosomal or genetic abnormalities
* CRL >84mm at the time of randomization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only pregnant women
Enrollment: 40 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
reassurance | at the time of screening test
  women will be asked about three questions, with up to 35 point for each question. 1) are you reassured about the test? 2) are you sure the test is correct? 3) test give me certain reassurance about the syndrome of my child
Anxiety | at the time of screening test
  anxiety test assessed by State-Trait Anxiety Inventory (STAI)
Satisfaction of the pregnant women | 11-13 weeks of gestation
  women will be asked if retrospectively they are happy with the assigned screening test as post-test satisfaction questionnaire:
  * Not all applicable (5 points)
  * Hardly applicable (10 points)
  * Somewhat applicable (20 points)
  * Very much applicable (35 points)
False positive rate | 1 week after test
  False positive rate for any trosomy and for trisomy 21
Anxiety | at the time of screening test
  anxiety test assessed by The Pregnancy-Related Anxiety Questionnaire (PRAQ-R)

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Migliorini S, Saccone G, Silvestro F, Massaro G, Arduino B, D'Alessandro P, Petti MT, Paino JAC, Guida M, Locci M, Zullo F. First-trimester screening based on cell-free DNA vs combined screening: A randomized clinical trial on women's experience. Prenat Diagn. 2020 Oct;40(11):1482-1488. doi: 10.1002/pd.5800. Epub 2020 Aug 13. PMID 32683755